CLINICAL TRIAL: NCT04432974
Title: Automatic Control of Total Intravenous Anesthesia: Closed-loop Delivery of Propofol and Remifentanil Using Bispectral Index as Feedback Variable
Brief Title: Automatic Control of Total Intravenous Anesthesia (ACTIVA)
Acronym: ACTIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Massimiliano Paltenghi, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-2861
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-06

CONDITIONS: Anesthesia
Keywords: Closed-loop Anesthesia; PID Control; Medical Control Systems; Automated Drug Delivery; Propofol; Remifentanil; Bispectral index; BIS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACTIVA (Experimental): ACTIVA closed-loop anesthesia control system
  Interventions: Device: Automatic closed-loop anesthesia

INTERVENTIONS:
Device: Automatic closed-loop anesthesia — Total intravenous anesthesia performed with the ACTIVA automatic control system
  Other Names: ACTIVA

SUMMARY:
This study concerns the clinical evaluation of a closed loop control system for the automatic administration of anesthetic drugs in TIVA (Total Intra Venous Anesthesia).

The purpose of the experimentation is to demonstrate that the control system under study is reliable, safe, applicable and capable of inducing and maintaining an optimal anesthetic level.

DETAILED DESCRIPTION:
This clinical study consists of the application of the ACTIVA control software for the infusion of intravenous drugs during general anesthesia according to the principle of closed-loop anesthesia.

The objective of the experimentation is to evaluate the reliability, safety and applicability of the infusion system for anesthetic drugs controlled by the ACTIVA software and to carry out the clinical evaluation of the automatic control system during the induction and maintenance of general intravenous anesthesia. The benefits for enrolled patients could be linked to greater stability of anesthesia in the induction and maintenance phases. Constant closed-loop control of infusions and the level of hypnosis could also reduce the hemodynamic impact that general anesthesia has on the patient, by reducing the onset of hypotension episodes.

Enrolled patients will undergo closed-loop anesthesia under the constant supervision of the investigator. The anesthetic drugs used are those recommended for general intravenous anesthesia: propofol and remifentanil.

Identification and description of the medical device:

The medical device object of the clinical investigation consists of the ACTIVA control software developed to control the infusion of anesthetic drugs during general intravenous anesthesia. ACTIVA software has been developed to optimize the infusion of anesthetic drugs according to a closed-loop system that allows the induction and maintenance of a constant and optimal level of anesthesia on the patient. ACTIVA control software is installed on a personal computer (PC).

The level of anesthesia is measured according to the Bispectral Index (BIS) which measures the depth of hypnosis. Through the measurement of the BIS, the administration of anesthetic drugs is automatically regulated by the ACTIVA software and constantly supervised by the anesthesiologist through the graphic interface integrated in the software.

The population for which the device is intended is made up of patients to undergo surgery for which general anesthesia is required, and intravenous anesthesia may be advantageous.

During its operation, the ACTIVA software maintains the desired BIS level, selected by the anesthesiologist through the graphical user interface, communicating the appropriate infusion rate of the propofol and remifentanil anesthetic drugs to the syringe pumps. ACTIVA software communicates with the pumps and the BIS monitoring system with serial connections. These connections are native to the instrumentation used; therefore, no type of modification or manipulation has been made on the medical devices used.

Closed-loop anesthesia:

A closed-loop system can be defined as an automatic control system that bases its operation on the principle of feedback. Its key elements are a system to be controlled, a measuring device (sensor), a controller and an actuator. The sensor measures the controlled variable (system output), which is compared with the desired set-point. The difference between the latter and the output, defined as an error, is used to calculate the value of the control variable (system input).

In the case of closed-loop anesthesia, the system to be controlled identifies with the patient, the actuator is represented by the syringe pump, the controlled variable corresponds to the BIS and the control variable is represented by the rate of infusion of the drugs.

The controller used is a proportional-integral-derivative (PID) it relates the error signal and the control variable by means of three constants (Kp, Ti and Td) allowing a correct infusion of the drugs considering the present value of the error ( proportional action), the past values of the error (integral action) and the advance of the future values of the error (derivative action). These three constants, if properly calibrated, allow to obtain a controller with good performance and robustness. For the ACTIVA system the calibration of these constants was carried out by means of optimization methods performed in simulation.

The anesthesiologist has at his disposal a PC with a graphical user interface through which he can control the start and end of the drug infusion and on which there are the commands through which it is possible to interact with the system. The graphical interface also reports indicators concerning the correct functioning of the control system. In case of malfunction of the ACTIVA software, the patient monitoring systems are never altered or damaged and the infusive pumps continue to operate in manual mode. Switching to manual control is always possible if the anesthesiologist considers it appropriate, even without the presence of system malfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing total intravenous general anesthesia for elective surgery

Exclusion Criteria:

* Patients under the age of 18
* Patients incapable of giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Paltenghi, MD, Principal Investigator — Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Locations (1):
- Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padula F, Ionescu C, Latronico N, Paltenghi M, Visioli A, Vivacqua G. Optimized PID control of depth of hypnosis in anesthesia. Comput Methods Programs Biomed. 2017 Jun;144:21-35. doi: 10.1016/j.cmpb.2017.03.013. Epub 2017 Mar 18. PMID 28495004
- [Background] Merigo L, Beschi M, Padula F, Latronico N, Paltenghi M, Visioli A. Event-Based control of depth of hypnosis in anesthesia. Comput Methods Programs Biomed. 2017 Aug;147:63-83. doi: 10.1016/j.cmpb.2017.06.007. Epub 2017 Jun 23. PMID 28734531
- [Derived] Schiavo M, Paltenghi M, Visioli A, Latronico N. Clinical Performance of a Bispectral Index Controlled Closed-Loop Administration System for Simultaneous Administration of Propofol and Remifentanil. Anesth Analg. 2025 May 1;140(5):1236-1238. doi: 10.1213/ANE.0000000000007289. No abstract available. PMID 39413036

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruited patients were patients scheduled for elective plastic surgery for whom general anesthesia performed in TIVA was deemed appropriate. The recruitments took place at the Spedali Civili di Brescia hospital, in the plastic surgery operating room.
  The first participant was enrolled on July 2, 2019 and the last participant was enrolled on April 4, 2023.
Pre-assignment Details: Patients were approached and informed of the possibility to participate in the study during the preoperative anesthesia visit, which takes place two weeks before the scheduled surgical procedure. If the patient wishes to participate in the study, the informed consent is obtained on the day of surgery, at the patient's arrival in the preoperative holding area.
Groups:
- ACTIVA: Participants received total intravenous anesthesia performed with the ACTIVA automatic control system.
Period: Overall Study
Arm/Group | ACTIVA
Started | 139
Operating Room Admission | 139
Operating Room Discharge | 139
Recovery Room Admission | 139
Recovery Room Discharge | 139
Ward 6 Hours Post-surgery | 139
Ward 24 Hours Post-surgery | 139
Completed | 139
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [46 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 139
Weight [Median (Inter-Quartile Range); unit: kg] | 70 [59 to 82]
Height [Median (Inter-Quartile Range); unit: cm] | 165 [160 to 171]
Mean arterial pressure [Median (Inter-Quartile Range); unit: mmHg] — Mean arterial pressure (MAP) is defined as diastolic pressure + 1/3(systolic pressure - diastolic pressure). It is non-invasively measured with an inflatable cuff by an electronic sphygmomanometer embedded in a multiparametric patient monitor at operating room admission, immediately before anesthesia.
  mmHg | 100 [96 to 122]
Heart rate [Median (Inter-Quartile Range); unit: beats per minute] — Heart rate measured at operating room admission, immediately before anesthesia.
  beats per minute | 71 [61 to 82]
ASA status [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) physical status classification system. ASA 1 = healthy person; ASA 2 = mild systemic disease; ASA 3 = severe systemic disease.
  Participants
    ASA 1 | 12
    ASA 2 | 96
    ASA 3 | 31
PONV risk [Count of Participants; unit: Participants] — Postoperative Nausea and Vomiting (PONV) risk according to the Apfel Simplified Risk Score: 0 (low risk) to 4 (high risk).
  Participants
    0 | 8
    1 | 34
    2 | 39
    3 | 45
    4 | 13
Type of surgery [Count of Participants; unit: Participants]
  Skin cancer exeresis | 54
  Mastectomy | 34
  Mastoplasty | 28
  Surgical treatment of wounds | 7
  Electrochemotherapy | 7
  Lipofilling | 5
  Eyelid surgery | 2
  Rhinoplasty | 1
  Brachioplasty | 1

OUTCOME MEASURES:

1. Primary Outcome: Depth of Hypnosis Adequacy
Description: The depth of hypnosis adequacy is assessed by evaluating, for each patient enrolled, the percentage of maintenance duration during which the Bispectral Index Scale (BIS) is kept within the recommended range from 40 to 60 (BIS [40,60]).
  The outcome measure is defined as the median of these percentages calculated over all the patients enrolled in the study.
  The median of the percentages, calculated over all the patients enrolled in the study, of the anesthesia maintenance duration in which the BIS is kept below 40 (BIS<40) is also specified.
  Maintenance duration is the period of time that goes from the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
  The BIS ranges from 0 (absence of brain activity) to 100 (fully awake patient).
Time Frame: During anesthesia from the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds to the point at which the automatic control is turned off (maintenance duration), an average of 2 hours.
Measure: Median (Inter-Quartile Range); unit: percentage of maintenance duration
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
percentage of maintenance duration
  BIS [40,60] | 79.4 [68.6 to 87.1]
  BIS<40 | 16.2 [10.0 to 26.2]

2. Secondary Outcome: Number of Participants for Which the System Showed Dysfunctions
Description: Number of participants for which the ACTIVA system showed dysfunctions. The results are presented in a table where each row indicates the type of dysfunction and the number of participants for which that particular type of dysfunction occurred.
Time Frame: During anesthesia from the time instant when the automatic control is started to the point at which the automatic control is turned off at the conclusion of surgery, an average of 2 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
Participants
  Venous access occlusion | 8
  Infusion pumps failure | 8
  No system dysfunctions | 123

3. Secondary Outcome: Levels of Satisfaction of the Experimenter Expressed as Number of Participants Who Have Received a Specific Score
Description: Levels of satisfaction of the experimenter regarding three aspects of the ACTIVA system.
  The first aspect is the ease of use of the ACTIVA software and its infusion system.
  The second aspect is the behavior of the ACTIVA system during the induction phase of anesthesia.
  The third aspect is the behavior of the ACTIVA system during the maintenance phase of anesthesia.
  For each aspect, the level of satisfaction is expressed by the experimenter by assigning a score on a scale ranging from 0 (extremely unsatisfied) to 10 (extremely satisfied).
  Thus, higher values represent a better outcome. Note that the scoring scale employed is the same for each of the three aspects. The results are reported in a table divided in three rows, one for each aspect evaluated.
  Each row is divided in eleven categories representing the scores from 0 to 10. For each category it is indicated the number of patients for which the experimenter expressed that specific score.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
Participants
  General level of satisfaction: 0 | 0
  General level of satisfaction: 1 | 0
  General level of satisfaction: 2 | 0
  General level of satisfaction: 3 | 0
  General level of satisfaction: 4 | 0
  General level of satisfaction: 5 | 0
  General level of satisfaction: 6 | 6
  General level of satisfaction: 7 | 23
  General level of satisfaction: 8 | 56
  General level of satisfaction: 9 | 42
  General level of satisfaction: 10 | 12
  Level of satisfaction regarding anesthesia induction: 0 | 0
  Level of satisfaction regarding anesthesia induction: 1 | 0
  Level of satisfaction regarding anesthesia induction: 2 | 0
  Level of satisfaction regarding anesthesia induction: 3 | 0
  Level of satisfaction regarding anesthesia induction: 4 | 0
  Level of satisfaction regarding anesthesia induction: 5 | 0
  Level of satisfaction regarding anesthesia induction: 6 | 7
  Level of satisfaction regarding anesthesia induction: 7 | 14
  Level of satisfaction regarding anesthesia induction: 8 | 35
  Level of satisfaction regarding anesthesia induction: 9 | 53
  Level of satisfaction regarding anesthesia induction: 10 | 30
  Level of satisfaction regarding anesthesia maintenance: 0 | 0
  Level of satisfaction regarding anesthesia maintenance: 1 | 0
  Level of satisfaction regarding anesthesia maintenance: 2 | 0
  Level of satisfaction regarding anesthesia maintenance: 3 | 0
  Level of satisfaction regarding anesthesia maintenance: 4 | 0
  Level of satisfaction regarding anesthesia maintenance: 5 | 0
  Level of satisfaction regarding anesthesia maintenance: 6 | 10
  Level of satisfaction regarding anesthesia maintenance: 7 | 16
  Level of satisfaction regarding anesthesia maintenance: 8 | 32
  Level of satisfaction regarding anesthesia maintenance: 9 | 48
  Level of satisfaction regarding anesthesia maintenance: 10 | 33

4. Secondary Outcome: Effect of Drugs Delivery on Heart Rate
Description: The effect of drugs delivery on heart rate is assessed by evaluating, for each patient enrolled, the percentage of the anesthesia maintenance duration in which the heart rate (HR) is kept inside the range from 50 to 100 beats per minute (HR [50,100]).
  The outcome measure is defined as the median of these percentages calculated over all the patients enrolled in the study.
  The median of the percentages, calculated over all the patients enrolled in the study, of the anesthesia maintenance duration in which the HR is kept below 50 (HR<50) is also specified.
  Maintenance duration is the period of time that goes from the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of maintanance duration
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
percentage of maintanance duration
  HR [50,100] | 99.7 [91.9 to 100.0]
  HR<50 | 0.3 [0.0 to 8.1]

5. Secondary Outcome: Effect of Drugs Delivery on Mean Arterial Pressure (MAP)
Description: The effect of drugs delivery on mean arterial pressure (MAP) is assessed by evaluating, for each patient enrolled, the anesthesia maintenance duration in which the non-invasively measured MAP is kept inside the range from 65 to 110 mmHg (MAP [65,110]).
  The outcome measure is defined as the median of these percentages calculated over all the patients enrolled in the study.
  The median of the percentages, calculated over all the patients enrolled in the study, of the anesthesia maintenance duration in which the MAP is kept below 65 (MAP<65) is also specified.
  Maintenance duration is the period of time that goes from the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
  MAP is defined as diastolic pressure + 1/3(systolic pressure - diastolic pressure).
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of maintenance duration
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
percentage of maintenance duration
  MAP [65,110] | 79.0 [63.1 to 92.1]
  MAP<65 | 15.7 [5.9 to 34.6]

6. Secondary Outcome: Postoperative Heart Rate Stability
Description: The postoperative heart rate is assessed by measuring the heart rate in beats per minute (bpm).
Time Frame: End of anesthesia (operating room discharge, recovery room admission, recovery room discharge), 6 hours after surgery, 24 hours after surgery.
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
beats per minute
  Operating room discharge | 72 [64 to 80]
  Recovery room admission | 74 [67 to 80]
  Recovery room discharge | 74 [65 to 80]
  6 hours after surgery | 74 [65 to 80]
  24 hours after surgery | 72 [68 to 80]

7. Secondary Outcome: Postoperative Mean Arterial Pressure (MAP) Stability
Description: The postoperative mean arterial pressure (MAP) stability is assessed by non-invasively measuring the MAP with an electronic sphygmomanometer trough an inflatable cuff.
  Mean arterial pressure (MAP) is defined as diastolic pressure + 1/3(systolic pressure - diastolic pressure).
Time Frame: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
mmHg
  Operating room discharge | 82 [75 to 93]
  Recovery room admission | 83 [77 to 92]
  Recovery room discharge | 85 [78 to 92]
  6 hours after surgery | 90 [80 to 97]
  24 hours after surgery | 88 [80 to 97]

8. Secondary Outcome: Postoperative Sedation Expressed as Number of Participants Who Have Received a Specific Score
Description: The postoperative sedation is assessed by means of a Sedation Score scale. It is a 3 point scale from 0 (fully awake) to 3 (fully sedated)
Time Frame: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
Participants
  Recovery room admission: 0 | 97
  Recovery room admission: 1 | 40
  Recovery room admission: 2 | 2
  Recovery room admission: 3 | 0
  Recovery room discharge: 0 | 115
  Recovery room discharge: 1 | 24
  Recovery room discharge: 2 | 0
  Recovery room discharge: 3 | 0
  6 hours after surgery: 0 | 135
  6 hours after surgery: 1 | 4
  6 hours after surgery: 2 | 0
  6 hours after surgery: 3 | 0
  24 hours after surgery: 0 | 139
  24 hours after surgery: 1 | 0
  24 hours after surgery: 2 | 0
  24 hours after surgery: 3 | 0

9. Secondary Outcome: Postoperative Nausea and Vomiting (PONV) Expressed as Number of Participants Who Have Received a Specific Score
Description: Postoperative Nausea and Vomiting is assessed by means of the Bellville PONV scale. It is a 3 point scale from 0 (no nausea & vomiting) to 3 (vomiting present)
Time Frame: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
Participants
  Recovery room admission: 0 | 136
  Recovery room admission: 1 | 3
  Recovery room admission: 2 | 0
  Recovery room admission: 3 | 0
  Recovery room discharge: 0 | 133
  Recovery room discharge: 1 | 4
  Recovery room discharge: 2 | 1
  Recovery room discharge: 3 | 1
  6 hours after surgery: 0 | 135
  6 hours after surgery: 1 | 4
  6 hours after surgery: 2 | 0
  6 hours after surgery: 3 | 0
  24 hours after surgery: 0 | 136
  24 hours after surgery: 1 | 2
  24 hours after surgery: 2 | 0
  24 hours after surgery: 3 | 1

10. Secondary Outcome: Postoperative Analgesia Expressed as Number of Participants Who Have Received a Specific Score
Description: The postoperative analgesia is assessed using a 10-point numeric rating scale (NRS). It is a 10 point scale from 0 (no pain) to 10 (maximum pain).
Time Frame: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
Participants
  Recovery room admission: 0 | 92
  Recovery room admission: 1 | 4
  Recovery room admission: 2 | 7
  Recovery room admission: 3 | 6
  Recovery room admission: 4 | 13
  Recovery room admission: 5 | 6
  Recovery room admission: 6 | 3
  Recovery room admission: 7 | 5
  Recovery room admission: 8 | 2
  Recovery room admission: 9 | 0
  Recovery room admission: 10 | 1
  Recovery room discharge: 0 | 74
  Recovery room discharge: 1 | 6
  Recovery room discharge: 2 | 16
  Recovery room discharge: 3 | 18
  Recovery room discharge: 4 | 7
  Recovery room discharge: 5 | 6
  Recovery room discharge: 6 | 5
  Recovery room discharge: 7 | 6
  Recovery room discharge: 8 | 1
  Recovery room discharge: 9 | 0
  Recovery room discharge: 10 | 0
  6 hours after surgery: 0 | 71
  6 hours after surgery: 1 | 12
  6 hours after surgery: 2 | 17
  6 hours after surgery: 3 | 18
  6 hours after surgery: 4 | 12
  6 hours after surgery: 5 | 4
  6 hours after surgery: 6 | 3
  6 hours after surgery: 7 | 2
  6 hours after surgery: 8 | 0
  6 hours after surgery: 9 | 0
  6 hours after surgery: 10 | 0
  24 hours after surgery: 0 | 88
  24 hours after surgery: 1 | 18
  24 hours after surgery: 2 | 12
  24 hours after surgery: 3 | 9
  24 hours after surgery: 4 | 7
  24 hours after surgery: 5 | 4
  24 hours after surgery: 6 | 0
  24 hours after surgery: 7 | 0
  24 hours after surgery: 8 | 1
  24 hours after surgery: 9 | 0
  24 hours after surgery: 10 | 0

11. Post Hoc Outcome: Induction Time
Description: The induction time is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
Time Frame: During anesthesia from the time instant when the automatic control is started to the point at which the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds, an average of 110 seconds.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
seconds | 103 [79 to 162]

12. Post Hoc Outcome: Lowest Bispectral Index (BIS) Induction
Description: The lowest Bispectral Index (BIS) is the lowest BIS value observed within the 60 seconds following the induction time.
  The BIS quantifies the cerebral activity and ranges from 99 (corresponding to a fully awake and aware patient) to 0 (corresponding to the absence of brain activity.
  For general anesthesia it is recommended to keep the BIS inside the range 40-60.
  Values above 60 represent a too light anesthesia while values below 40 represents a too deep anesthesia.
Time Frame: During anesthesia from the time instant when the automatic control is started to 60 seconds following the induction time, an average of 170 seconds.
Measure: Median (Inter-Quartile Range); unit: units on a scale (BIS)
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
units on a scale (BIS) | 42 [36 to 45]

13. Post Hoc Outcome: Propofol Induction Dose
Description: Propofol dose administered by the system throughout the induction time.
Time Frame: During anesthesia from the time instant when the automatic control is started to the point at which the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds, an average of 170 seconds.
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
mg/kg | 1.90 [1.63 to 2.19]

14. Post Hoc Outcome: Remifentanil Induction Dose
Description: Remifentanil dose administered by the system throughout the induction time.
Time Frame: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ug/kg
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
ug/kg | 2.16 [1.73 to 2.61]

15. Post Hoc Outcome: Lowest Heart Rate Induction
Description: The lowest heart rate is the lowest heart rate value observed within the 5 minutes following the induction time.
Time Frame: During anesthesia from the time instant when the automatic control is started to the 5 minutes following the induction time, an average of 410 seconds.
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
beats per minute | 54 [48 to 59]

16. Post Hoc Outcome: Lowest Mean Arterial Pressure (MAP) Induction
Description: The lowest mean arterial pressure (MAP) is the lowest value of the MAP observed within the 5 minutes following the induction time.
  It is assessed by non-invasively measuring the MAP with an electronic sphygmomanometer embedded in a multiparametric patient monitor through an inflatable cuff.
  Mean arterial pressure (MAP) is defined as diastolic pressure + 1/3(systolic pressure - diastolic pressure).
Time Frame: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
mmHg | 69 [58 to 76]

17. Post Hoc Outcome: Number of Participants With Burst-Suppression Episode Following Anesthesia Induction
Description: Number of Participants that showed the occurrence of a burst-suppression episode within the 5 minutes following the induction time.
  A burst-suppression episode is defined as a value of burst-suppression ratio (BSR) above 10% for at least 60 seconds.
Time Frame: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
Participants | 6

18. Post Hoc Outcome: MDPE
Description: The MDPE is the median performance error calculated during the maintenance phase. The performance error (PE) is calculated for each patient (i) and for each BIS sample (j) according to the formula: PEij=((BISij-BIS_Target)/BIS_Target)*100, where BIS_Target is set equal to 50.
  The MDPE is a measure of bias and describes whether the measured BIS values are systematically distributed either above or below the BIS target.
  The MDPE is calculated according to the formula: MDPEi=median{PEij}. The maintenance phase is defined as the period of time that goes from the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of target BIS value
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
percentage of target BIS value | -10 [-16 to -6]

19. Post Hoc Outcome: MDAPE
Description: The MDAPE is the median absolute performance error calculated during the maintenance phase. The performance error (PE) is calculated for each patient (i) and for each BIS sample (j) according to the formula: PEij=((BISij-BIS_Target)/BIS_Target)*100, where BIS_Target is set equal to 50.
  The MDAPE is a measure of inaccuracy. The MDAPE is calculated according to the formula: MDAPEi=median{|PEij|}. The maintenance phase is defined as the period of time that goes from the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of target BIS value
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
percentage of target BIS value | 12 [10 to 16]

20. Post Hoc Outcome: WOBBLE
Description: The WOBBLE is an index of time-related changes in the performance and measures the intra-patient variability in performance errors.
  It is calculated during the maintenance phase. The performance error (PE) is calculated for each patient (i) and for each BIS sample (j) according to the formula: PEij=((BISij BIS_Target)/BIS_Target)*100, where BIS_Target is set equal to 50.
  The WOBBLE is calculated according to the formula: WOBBLEi=median{|PEij-MDPEi|}.
  The maintenance phase is defined as the period of time that goes from the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of target BIS value
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
percentage of target BIS value | 8 [6 to 10]

21. Post Hoc Outcome: Global Score (GS)
Description: The Global Score (GS) is a performance index that characterize the overall control performance.
  It is calculated as (MDAPE+WOBBLE)/BIS [40,60].
  For each patient (i) and for each Bispectral Index Scale (BIS) sample (j):
  PEij=((BISij BIS_Target)/BIS_Target)*100, with BIS_Target=50. MDAPEi=median{|PEij|}. WOBBLEi=median{|PEij-MDPEi|}. BIS [40,60] is the percentage of the anesthesia maintenance duration in which the BIS is kept between 40 and 60.
  The maintenance phase is defined as the period of time that goes from the end of anesthesia induction, defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds, to the point at which the automatic control is turned off at the conclusion of surgery.
  The GS ranges from zero to infinity. The lower the GS, the better the control performance. Specifically, a GS value of zero would correspond to the case where the BIS is always maintained at its target value.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Dimensionless
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
Dimensionless | 26.3 [22.2 to 36.7]

22. Post Hoc Outcome: Median Maintenance Propofol Infusion Rate
Description: It is the median value of the propofol infusion rate administered by the ACTIVA system during the maintenance phase of anesthesia.
  The outcome measure is defined as the median of the propofol infusion rates administered by the ACTIVA system during the maintenance phase of anesthesia calculated over all the patients enrolled in the study.
  The maintenance phase is defined as the period of time that goes from the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg/kg/h
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
mg/kg/h | 6.19 [5.05 to 7.26]

23. Post Hoc Outcome: Median Maintenance Remifentanil Infusion Rate
Description: It is the median value of the remifentanil infusion rate administered by the ACTIVA system during the maintenance phase of anesthesia.
  The outcome measure is defined as the median of the remifentanil infusion rates administered by the ACTIVA system during the maintenance phase of anesthesia calculated over all the patients enrolled in the study.
  The maintenance phase is defined as the period of time that goes from the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ug/kg/min
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
ug/kg/min | 0.16 [0.13 to 0.21]

24. Post Hoc Outcome: Median Maintenance Propofol Effect-Site Concentration
Description: It is the median propofol effect-site concentration achieved by the ACTIVA system during the maintenance phase of anesthesia.
  It is estimated according to the Schnider model. The outcome measure is defined as the median of the propofol effect-site concentrations achieved by the ACTIVA system during the maintenance phase of anesthesia calculated over all the patients enrolled in the study.
  The maintenance phase is defined as the period of time that goes from the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
ug/ml | 2.72 [2.41 to 3.18]

25. Post Hoc Outcome: Median Maintenance Remifentanil Effect-Site Concentration
Description: It is the median remifentanil effect-site concentration achieved by the ACTIVA system during the maintenance phase of anesthesia.
  It is estimated according to the Minto model. The outcome measure is defined as the median of the remifentanil effect-site concentrations achieved by the ACTIVA system during the maintenance phase of anesthesia calculated over all the patients enrolled in the study.
  The maintenance phase is defined as the period of time that goes from the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
ng/ml | 5.02 [4.21 to 6.25]

26. Post Hoc Outcome: Number of Participants With Burst-Suppression Episode During Anesthesia Maintenance
Description: Number of Participants that showed the occurrence of a burst-suppression episode during the maintenance phase.
  A burst-suppression episode is defined as a value of burst-suppression ratio (BSR) above 10% for at least 60 seconds.
  The maintenance phase here is defined as the period of time that goes from the 5 minutes after the end of anesthesia induction to the point at which the automatic control is turned off at the conclusion of surgery.
  The end of anesthesia induction is defined as the time instant when the BIS drops below 60 for the first time and remains there for the subsequent 30 seconds.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
Participants | 25

27. Post Hoc Outcome: Number of Participants That Received Hemodynamic Interventions
Description: Number of Participants that showed cases of hypotension treated with ephedrine or etilefrine before and after the beginning of the surgical stimulation (incision).
Time Frame: During anesthesia from the time instant when the automatic control is started to incision for the cases before incision. During anesthesia from incision to the time instant when the automatic control is stopped for the cases after incision.
Measure: Count of Participants; unit: Participants
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
Participants
  Before incision | 26
  After incision | 71

28. Post Hoc Outcome: Extubation Time
Description: The extubation time is the time interval that elapses from the time instant when the automatic control is stopped to when the patient is extubated.
  It is an indicator of the awakening time.
Time Frame: During anesthesia from the time instant when the automatic control is stopped to when the patient is extubated, up to 11 minutes.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | ACTIVA
Number analyzed (Participants) | 139
seconds | 496 [374 to 608]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Adverse events are noted as soon as they occur by the prinipal investigator on the data collection form of each patient enrolled in the study.
Arm/Group | ACTIVA
All-Cause Mortality (participants affected / at risk) | 0/139
Serious Adverse Events (participants affected / at risk) | 0/139
Other Adverse Events (participants affected / at risk) | 0/139

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT04432974/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT04432974/SAP_001.pdf